CLINICAL TRIAL: NCT02554604
Title: Identifying HDL Composition and Function in Preeclamptic and Normal Pregnancies and Volatile Organic Compounds in Maternal Saliva Characteristic of Preeclampsia
Brief Title: Identifying HDL Composition and Function in Preeclamptic and Normal Pregnancies
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, yael einbinder, Staff Nephrologist, Meir Medical Center
Other Study IDs: 0122-15
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2018-08

CONDITIONS: HDL Cholesterol; Preeclampsia; Saliva
Keywords: HDL; Preeclampsia; saliva
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant woman: Pregnant woman with identified risk factors for the development of preeclampsia

SUMMARY:
The study is design to assess if there is a correlation between diagnosis of preeclampsia and its severity to changes in HDL quality, in terms of composition and function and to determine whether preeclampsia-induced changes in VOCs in saliva can be used for the early diagnosis of preeclampsia.

DETAILED DESCRIPTION:
Scientific background Preeclampsia is a syndrome characterized by the onset of hypertension and proteinuria or other end-organ dysfunction. It develops after 20 weeks of gestation and can cause significant maternal and fetal morbidity and mortality (1,2). The pathophysiology of preeclampsia is thought to be developmental abnormalities of placental vasculature leading to placental under-perfusion or ischemia. This ischemia is believed to mediate the release of anti-angiogenic factors into the maternal circulation, causing endothelial dysfunction, hypertension and end-organ injury (2). The elemental factor that leads to the development of placental vasculature abnormalities is still to be elucidated. However, histological changes in the placenta include atherosis (lipid laden cells in the wall of the arteriole), fibrinoid necrosis, thrombosis, sclerotic narrowing of arterioles, and placental infarction, all of which are similar to findings seen in atherosclerotic plaque (1-3). Another close association between the mechanisms of preeclampsia and atherosclerosis was found in large epidemiological studies that demonstrated a strong correlation between preeclampsia (PET) and the development of cardiovascular disease later in life (4). Women with PET are more likely than those with normal pregnancy to develop chronic hypertension, cardiovascular disease, stroke, diabetes and end-stage renal disease (1,4).Common atherosclerotic diseases, such as hypertension, chronic kidney disease (CKD), hypercholesterolemia and diabetes are strongly associated with preeclampsia during pregnancy (5-6).

Large epidemiologic and experimental studies have shown an association between low levels of high density lipids (HDL) in the blood and increased cardiovascular risk (7). The cardioprotective properties of HDL are thought to be composed of several mechanisms, including regulation of endothelial functions that enhance NO production and maintaining endothelial integrity, as well as anti-inflammatory, anti-oxidative and anti-thrombotic effects (8-9). However, pharmacological studies reported that increases in plasma HDL did not improve cardiovascular outcomes (10-12).

At the same time, emerging data have revealed the importance of the quality of the HDL more than its quantity. HDL from patients with CKD was found to lose its anti-atherogenic and endothelial protective effects. In a study by Shroff et al. (13), HDL from patients with CKD was incubated with a primary endothelial cell line. Several endothelial functions, such as reduced NO production, permission of SO production, increased VCAM-1 expression and reduction of cholesterol efflux capacity were decreased compared to those of HDL from healthy individuals. These effects were associated with vascular dysfunction markers in those patients, such as high levels of urate, angiopoeitin and IL-6, as well as poor vascular function measurements, as measured by aortic pulse velocity and carotid intima media thickness. These negative functions increased as CKD severity progressed and showed a partial improvement after kidney transplantation (13).

Information regarding the composition and function of serum lipids and lipoproteins among preeclamptic pregnancies compared to normal pregnancies is scarce. Early pregnancy dyslipidemia, particularly hypertriglyceridemia appears to be associated with increased risk of preeclampsia (14). However, equivocal results were found regarding paraoxonase 1 (PON1) activity, which is an antioxidative enzyme found in HDL that inhibits low density lipid (LDL) and HDL oxidation. PON1 activity is decreased in diseases associated with endothelial activation and dysfunction including diabetes, hypercholesterolemia and cardiovascular disease (15). Demir et al. (16) found low levels of HDL, ApoA1 and paraoxonase activity in preeclamptic compared to normal pregnancies, whereas Acikgoz et al. (17) demonstrated significantly higher PON1 activity in preeclamptic compared to normal pregnancies.

Saliva contains constituents that reflect a diseased or physiologic state of the human body and hence could be utilized for diagnostic purposes. The sources and composition of whole saliva (oral fluid) are unique and complex. Saliva consists of secretions from salivary glands and gingival crevicular fluid, oral mucosa transudate, secretions from nasal and pharyngeal mucosa, nonadherent bacteria, desquamated oral epithelial cells, keratin debris, blood cells, and possibly food or medication residuals (18). Its functions include lubrication, digestion, antimicrobial activity, facilitating remineralization of dental enamel, and maintaining normal taste sensation (19). These important functions are achieved by the various chemical components of saliva including water, inorganic compounds (ions), organic compounds (non-proteins and lipids), protein/polypeptides, and hormones (19). The search for reliable salivary biomarkers has developed rapidly, especially in oral cancers, spurred by the fact that collecting saliva is simpler and less invasive than drawing blood.

Salvador-Moysén et al. (20) aimed to determine the usefulness of salivary cortisol as a predictor of preeclampsia in adolescents. They found that cortisol concentrations >14.9 nmol/L were observed in the group that developed preeclampsia, whereas the control group had values <10.1 nmol/L.

Volatile organic compounds (VOC) can be detected in the breath and blood and used for the early detection and characterization of the development and progression of diseases (21). Many of the VOC that are detected in the breath are systemic or endogenous and are produced during physiological processes, but the metabolic routes behind their production are known for only a few (22). Other VOCs are exogenous and result from external contamination through inhaled air or ingested foods or drinks.

Solid phase microextraction (SPME) is a simple, automated, rapid technique for VOC detection combined with gas chromatography-mass spectrometry (GC-MS) (20). To the best of our knowledge, no studies have been conducted to identify VOC in saliva from preeclamptic women.

Objectives

1. There is a correlation between diagnosis of preeclampsia and its severity to changes in HDL quality, in terms of composition and function.
2. Determine whether preeclampsia-induced changes in VOCs in saliva can be used for the early diagnosis of preeclampsia.

Research goals

1. Assess:

   HDL composition and function of normal and preeclamptic pregnancies at weeks 12-14 (second trimester), weeks 28-30 (third trimester) and at delivery Apo-A1 properties, PON1 activity HDL size HDL lipid content HDL antioxidant activity (toward LDL and macrophages) HDL-mediated cholesterol efflux from macrophages
2. Evaluate the effects of HDL from women with PET, normal pregnancies and non-pregnant women, on primary endothelial culture regarding proteins, mRNA and miRNAs, which are significant components in normal endothelial function and related to inflammatory response.
3. Evaluate differences in the genomic and lipid profiles of cord blood and placentas from women with PET, normal pregnancies and non-pregnant women
4. Identify VOC in saliva, as early biomarkers of PET during the second and third trimesters and at delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman followed in Community Obstetric Clinics and in the High Risk Obstetric Clinic at Meir Medical Center who agree to participate in the study.
* Woman will be recruited based on the presence of one or more risk factors for the development of preeclampsia including: first pregnancy, overweight at the beginning of pregnancy or significant weight gain during pregnancy , previous history of preeclampsia and a first degree family member with a history of preeclampsia.

Exclusion Criteria:

* Participants with multiple fetuses (previous medical history of hypertension, chronic kidney disease, diabetes mellitus) or who are unable to provide informed consent due to language barrier or other cause, will be excluded from the study.
* Patients who were not recruited to the study at the beginning of pregnancy will be allowed to join at any stage, including on delivery day.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant woman followed in Community Obstetric Clinics and in the High Risk Obstetric Clinic at Meir Medical Center who agree to participate in the study.
  Woman will be recruited based on the presence of one or more risk factors for the development of preeclampsia including: first pregnancy, overweight at the beginning of pregnancy or significant weight gain during pregnancy , previous history of preeclampsia and a first degree family member with a history of preeclampsia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
signs and symptoms of preeclampsia | 9 months
  blood pressure, BMI, presence of edema, urinalysis-proteinuria, in addition to all routine second and third trimester checkups that will be documented.

SECONDARY OUTCOMES:
Blood samples for lipid profile and HDL | 9 months
  blood samples will be collected from the volunteers during their pregnancy follow up during the first trimester 12-14 weeks, second trimester 28-32 weeks and on delivery day.

OTHER OUTCOMES:
Saliva measurement | 9 months
  Saliva samples will be collected from the volunteers during their pregnancy follow up during the first trimester 12-14 weeks, second trimester 28-32 weeks and on delivery day.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Dr. Yael Einbinder, Kfar Saba
  - Laboratory of Renal Physiology, Meir Medical Center ,, Kfar Saba

IPD SHARING:
Plan to Share IPD: No